CLINICAL TRIAL: NCT06827535
Title: Long-term Vascular, Functional and Morphological Changes in Glaucoma and Ocular Hypertensive Patients
Acronym: Ippocrate
Status: Enrolling by invitation | Type: Observational
Sponsor: Mario Stirpe (Other)
Responsible Party: Sponsor-Investigator, Mario Stirpe, Dr, Fondazione G.B. Bietti, IRCCS
Organization: Fondazione G.B. Bietti, IRCCS (Other)
Other Study IDs: GLC 04-24
Record Dates: First submitted 2025-01-30; First posted 2025-02-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma; ocular hypertension; vascular changes; morphological changes; functional changes
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Glaucoma: iagnosis of primary glaucoma (open or closed angle) or secondary glaucoma (pseudoexfoliative or pigmentary) defined by the presence of a glaucomatous defect of the optic nerve and/or a perimetric glaucomatous defect as defined by European guidelines
- Ocular Hypertension: Diagnosis of ocular hypertension (defined by the presence of intraocular pressure values ≥22 mmHg, optic nerve and visual field examination within normal limits).
- Healthy subjects: No optic nerve disease IOP < 21 mmHg

SUMMARY:
This is an observational study involving patients with glaucoma, those with ocular hypertension and healthy subjects.

The aim of the study is the long term evaluation of functional, vascular and morphological changes in glaucoma and ocular hypertensive patients, compared to healthy subjects, to analyze the temporal relationship of these changes.

DETAILED DESCRIPTION:
This is an observational study involving patients with glaucoma, those with ocular hypertension and healthy subjects.

The aim of the study is the long term evaluation of functional, vascular and morphological changes in glaucoma and ocular hypertensive patients, compared to healthy subjects, to analyze the temporal relationship of these changes.

Secondary aims of the study are:

* evaluating the effect of age on functional, morphological and vascular changes and their relationship,
* evaluating the effect of myopia on functional, morphological and vascular changes and their relationship,
* evaluating clinical and demographic factors associated with glaucoma onset and progression,
* evaluating the effects of vascular, functional and morphological changes on quality of life

During the study patients will undergo BCVA assessment, biomicroscopy, IOP measurement, CCT measurement, gonioscopy, visual field test, optic nerve head and macula OCT scan, OCT angiography scan, fundoscopy, every 6 months (for glaucoma and ocular hypertensive patients) and every 12 months (for healthy subjects). The study lasts 3 years.

Four Italian glaucoma center will partecipate in this study, in addition to the promoter.

Four hundred patients and 100 healthy subjects will be involved.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary glaucoma (open or closed angle) or secondary glaucoma (pseudoexfoliative or pigmentary) defined by the presence of a glaucomatous defect of the optic nerve and/or a perimetric glaucomatous defect as defined by the European guidelines
* Diagnosis of ocular hypertension (defined by the presence of intraocular pressure values≥22 mmHg, optic nerve and visual field examination within normal limits)
* No Optic nerve disease and IOP<21mmHg for healthy subjects
* Age>18 years
* Able to read and sing the informed consent form

Exclusion Criteria:

1. BCVA <5/10
2. Previous eye surgery, except glaucoma surgery or removal of cataracts performed more than 6 months prior to enrollment
3. Other pathologies that can cause alterations of the optic nerve or visual field defects
4. Presence of maculopathies
5. Inability to perform visual field tests
6. Opacity of the dioptric media such that it is not possible to perform reliable OCT and OCTA of acceptable quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People attending the hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-11-14 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Rate of disease progression | Up to 3 years
  Rate of progression of functional, morphological and vascular parameters, calculated on the basis of tests repeated over time

SECONDARY OUTCOMES:
Rate of disease progression in relation to age | Up to 3 years
  Rate of progression of functional, morphological and vascular parameters, in relation to age
Rate of disease progression in relation to myopia | Up to 3 years
  Rate of progression of functional, morphological and vascular parameters, in relation to myopia
Rate of disease progression in relation to demographic data | Up to 3 years
  Rate of progression of functional, morphological and vascular parameters, in relation to clinical and demographic factors collected at baseline (visual acuity, axial length, diagnosis, sex, stage of the disease, etc.)
Quality of life in glaucoma and ocular hypertensive patients | Up to 3 years
  Quality of life questionnaire (National Eye Institute Visual Function Questionnaire-25) scores over time.
  The minimum value is 0, the maximum value is 100. Higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Ospedale San Paolo - ASST Santi Paolo e Carlo, Milan, Italy
  - Ospedale Maggiore della Carità, Novara, Italy
  - Irccs-Fondazione Gb Bietti, Rome, Italy
  - Azienda Ospedaliera Universitaria di Sassari, Dipartimento di Medicina, Chirurgia e Farmacologia Università di Sassari, Sassari, Italy
  - Clinica Oculistica, DiNOGMI, Università di Genova, Genoa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sotimehin AE, Ramulu PY. Measuring Disability in Glaucoma. J Glaucoma. 2018 Nov;27(11):939-949. doi: 10.1097/IJG.0000000000001068. PMID 30161076
- [Background] Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002 Oct;120(10):1268-79. doi: 10.1001/archopht.120.10.1268. PMID 12365904